CLINICAL TRIAL: NCT02791464
Title: Transcendental Meditation and Reduced Trauma Symptoms in Women Inmates: A Randomized Controlled Pilot Study
Brief Title: Transcendental Meditation and Reduced Trauma Symptoms in Women Inmates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: Western Oregon University (Other); Maharishi University of Management Research Institute (Other)
Responsible Party: Principal Investigator, Sanford Nidich, Principal Investigator, Associate Director, Maharishi International University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DLF1008; NCT03232060 (obsolete NCT alias)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Meditation; TM; PTSD; Trauma; Female Prisoners
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- wait list control (No Intervention): Waitlist control subjects interested in learning the TM program will be asked to wait for 4 months before learning if they were randomly assigned to this comparison group. Controls will receive usual medical care during 4 month intervention period.
- Transcendental Meditation (Experimental): The TM technique is a simple, effortless, mental technique to reducing stress which allows the mind to experience finer levels of the thinking process to achieve a state of restful alertness. The Transcendental Meditation program will be taught as a standard seven-step program over five consecutive days.
  Interventions: Behavioral: Transcendental Meditation program

INTERVENTIONS:
Behavioral: Transcendental Meditation program — a mental technique using a mantra or 'soothing sound' that refines the thought process enabling the mind to 'transcend' its own thinking process and experience a state of pure consciousness. Subjects practice this technique twice a day for 20 minutes sitting in chair with eyes closed.
  Other Names: TM technique
  Arms: Transcendental Meditation

SUMMARY:
The pilot study investigates the potential benefits of the Transcendental Meditation program in reducing trauma, including PTSD, in female prisoners. Subjects will be randomly assigned to either the TM program or a wait list control group for a period of four months.

DETAILED DESCRIPTION:
This randomized controlled pilot study will evaluate the effects of Transcendental Meditation ® (TM) on female offenders with trauma. Twenty-two inmates at the Coffee Creek Correctional Facility in Wilsonville, Oregon, with at least four months left of incarceration, will be enrolled in the study. Subjects will be randomly assigned to either a TM (n=11) or a wait-list control group (n=11). Subjects will be measured at baseline and four-month posttest, using the Posttraumatic Stress Disorder Checklist-Civilian version (PCL-C) Twenty of the subjects (10 in each group) will take part in their treatment assignment and complete post-testing.

ELIGIBILITY:
Inclusion Criteria:

* female inmates, at least 4 months left of incarceration, signed written informed consent prior to baseline testing

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Checklist- Civilian Version (PCL-C) total score | 4 months
  The PCL-C is a widely-used 17-item self-report questionnaire of trauma symptom with total score and intrusions, avoidance and hyperarousal subscales

CONTACTS AND LOCATIONS:
Overall Officials: Fred Travis, PhD, Study Chair — Maharishi University of Management Research Institute

IPD SHARING:
Plan to Share IPD: Yes
inquiring investigators may contact the principal investigator, Dr Sanford Nidich, for data share plans. Database resides with the PI and the biostatistician